CLINICAL TRIAL: NCT03294148
Title: Mind-body Treatments for Chronic Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Radiological Society of North America (Other); National Institutes of Health (NIH) (NIH); Psychophysiologic Disorders Society (Other); Foundation for the Science of Therapeutic Encounter (Other)
Responsible Party: Principal Investigator, Jonathan Ashar, Graduate student under the supervision of PI Wager, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0544
Record Dates: First submitted 2017-09-13; First posted 2017-09-26 (Actual); Results first posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Chronic Pain; Back Pain Lower Back Chronic; Back Pain, Low
Keywords: Placebo; Back; Pain; Chronic; Mind-Body
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two different studies: a placebo vs. waitlist study or a psychotherapy vs. waitlist study, with randomization stratified on pain intensity, age, gender, and opioid use. After an eligibility session, eligible participants will be randomized to the treatment group or the waitlist group (with a ratio of 2:1 treatment:waitlist), using a computer-generated random sequence. This scheme will result in three equally sized groups-placebo, psychotherapy, and waitlist-as the investigators will collapse data from the waitlist arms in the two studies for analyses. The investigators do not use a standard three-way randomization because the investigators do not want placebo participants to think they are in a control condition. Thus, the investigators constrain participant's expectations to either injection vs. waitlist or to psychotherapy vs. waitlist.
Who Masked: Outcomes Assessor
Masking Description: Researchers will not know which treatment the participants will be receiving (placebo or psychotherapy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Experimental): The open-label placebo treatment the investigators will use is based on past open-label placebo trials (Kam-Hansen et al., 2014; Kaptchuk et al., 2010; Kelley et al., 2012). Prior to treatment administration, patients will view a brief (~3 min) video summarizing scientific findings regarding the therapeutic power of placebo treatments. The video will describe established findings regarding placebo and suggest that placebos may still work even when patients know the treatment is a placebo. The video will state that believing in the placebo is not necessary, and the investigators ask only that patients keep an open mind. Patients will then receive a subcutaneous injection of 1ml medical grade saline into the lower back. The injection will be administered near the location of the pain, as specified by the participant. The investigators will use a standard needle used in subcutaneous injections of 27 gauge with a length from 1in to 1.5in.
  Interventions: Other: Open-Label Placebo Treatment for Chronic Back Pain
- Psychotherapy (Experimental): Psychotherapy will consist of one initial medical history session with Co-I Schubiner, followed by twice weekly 50 minute psychotherapy sessions for 4 weeks with a therapist, for a total of 9 sessions maximum. The purpose of the initial medical history session is to help evaluate the likelihood that the patient's back pain is caused by structural conditions in the back. Dr. Schubiner will then speak with patients for a 1 hour session in which he collects their medical history and discusses different possible causes of their back pain with them. This session will be conducted by phone, by HIPAA-compliant Zoom, or by another HIPAA-compliant videoconferencing technology in consultation with the OIT team at Dr. Schubiner's hospital.
  Interventions: Behavioral: Psychotherapy Treatment for Chronic Back Pain
- Waitlist (No Intervention): Wait-listed patients will be asked not to change their treatment regime for the 4 weeks in between their two fMRI sessions. Wait-listed patients in the placebo injection arm will be offered the opportunity to receive the placebo treatment (optional). Waitlisted participants in the psychotherapy arm will be given a copy of Dr. Schubiner's book and free access to his online self-help program (optional to accept these).

INTERVENTIONS:
Other: Open-Label Placebo Treatment for Chronic Back Pain — Subcutaneous injection of 1ml medical grade saline into the lower back.
  Arms: Placebo
Behavioral: Psychotherapy Treatment for Chronic Back Pain — Twice weekly 50 minute psychotherapy sessions for 4 weeks, plus an initial medical history session
  Arms: Psychotherapy

SUMMARY:
Participants with chronic back pain will complete an online prescreen. They will then be randomized to one of two different studies: a placebo vs. waitlist study or a psychotherapy vs. waitlist study, with randomization stratified on pain intensity, age, gender, and opioid use. Participants will then complete an in-person eligibility session, and eligible participants will be scheduled for the baseline assessment session. Following the baseline assessment session, participants will then be randomized to the treatment group or the waitlist group (with a ratio of 2:1 treatment:waitlist), using a computer-generated random sequence.

This scheme will result in three equally sized groups-placebo, psychotherapy, and waitlist-as the investigators will collapse data from the waitlist arms in the two studies for analyses. The investigators do not use a standard three-way randomization because the investigators do not want placebo participants to think they are in a control condition. Thus, the investigators constrain participant's expectations to either injection vs. waitlist or to psychotherapy vs. waitlist.

The placebo treatment is a subcutaneous injection of saline into the back. Participants will know that the treatment is a placebo, i.e., it is an "open label" placebo. Psychotherapy (8 sessions) will be supervised by Alan Gordon and Howard Schubiner.

Functional MRI brain imaging, self-reported clinical outcomes, and behavioral measures will be collected pre- and post-treatment. A brief follow-up survey will be sent at months 1, 2, 3, 6, and 12 after the final assessment session. These will provide longer term data about the trajectory and durability of patient improvement.

Additionally, a group of healthy controls, with no history of back pain, will complete the baseline assessment. They will serve as a comparison group to probe whether the patterns of observed brain activity is specific to CBP patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 21 to 70 with CBP will be enrolled.
* CBP will be defined according to the criteria established by a recent NIH task force (Deyo et al., 2014). Pain duration must be at least 3 months, with back pain being an ongoing problem for at least half the days of the last 6 months. That is, patients can meet criteria by either reporting pain every day for the past 3 months, or by reporting pain on half or more of the days for the past 6+ months. This will be determined by asking patients: (1) How long has back pain has been an ongoing problem for you? (2) How often has low back pain been an ongoing problem for you over the past 6 months? A response of greater than 3 months to question 1 and a response of ''at least half the days in the past 6 months'' to question 2 would define CBP.
* Patients must rate pain intensity at 40/100 or greater on the Brief Pain Inventory-Short Form (BPI-SF), in keeping with inclusion criteria from previous CBP trials (Baliki et al., 2012; Cherkin et al., 2016; Hashmi et al., 2013; Seminowicz et al., 2011).
* Back pain must be elicited by our back pain device (see below).
* Participants must also be comfortable and able to communicate via email or text message, as several study measures are collected in this manner (see below).

Exclusion Criteria:

* Back pain associated with compensation or litigation issues as determined by self-report within the past year.
* Leg pain is greater than back pain. This suggests neuropathic pain, which may be less responsive to placebo or psychotherapy.
* Difficulty participating for technical/logistical issues (e.g., unable to get to assessment sessions).
* Self-reported diagnoses of schizophrenia, multiple personality disorder, or dissociative identity disorder.
* Self-reported use of intravenous drugs, due to concerns about infections and subject compliance with experimental protocols.
* Inability to undergo MRI as determined by MRI safety screen (e.g., pregnancy, metal in body, claustrophobia, using the standard screen conducted by the MRI imaging facility).
* Hypersensitive or hyposensitive to pressure pain: unable to tolerate 7kg/cm2 stimulation or reporting no pain for 4kg/cm2 stimulation; see further details below.
* Current regular use of an immunosuppressant drug, such as steroids. Such drugs interfere with immunoassay results.
* Self-reported history of metastasizing cancers-cancer of the breast, thyroid, lung, kidney, prostate or blood cancers.
* Self-reported history of stroke, brain surgery, or brain tumor.
* Self-reported diagnosis of a specific inflammatory disorder: rheumatoid arthritis, polymyalgia rheumatica, scleroderma, Lupus, or polymyositis.
* Unexplained, unintended weight loss of 20 lbs. or more in the past year.
* Cauda Equina syndrome, as screened for by self-reported inability to control bowel or bladder function.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2019-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tor Wager, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

REFERENCES:
- [Background] Annersten M, Willman A. Performing subcutaneous injections: a literature review. Worldviews Evid Based Nurs. 2005;2(3):122-30. doi: 10.1111/j.1741-6787.2005.00030.x. PMID 17040533
- [Background] Ashar YK, Chang LJ, Wager TD. Brain Mechanisms of the Placebo Effect: An Affective Appraisal Account. Annu Rev Clin Psychol. 2017 May 8;13:73-98. doi: 10.1146/annurev-clinpsy-021815-093015. Epub 2017 Mar 27. PMID 28375723
- [Background] Atlas LY, Bolger N, Lindquist MA, Wager TD. Brain mediators of predictive cue effects on perceived pain. J Neurosci. 2010 Sep 29;30(39):12964-77. doi: 10.1523/JNEUROSCI.0057-10.2010. PMID 20881115
- [Background] Baliki MN, Petre B, Torbey S, Herrmann KM, Huang L, Schnitzer TJ, Fields HL, Apkarian AV. Corticostriatal functional connectivity predicts transition to chronic back pain. Nat Neurosci. 2012 Jul 1;15(8):1117-9. doi: 10.1038/nn.3153. PMID 22751038
- [Background] Becker GM, DeGroot MH, Marschak J. Measuring utility by a single-response sequential method. Behav Sci. 1964 Jul;9(3):226-32. doi: 10.1002/bs.3830090304. No abstract available. PMID 5888778
- [Background] Bicket MC, Gupta A, Brown CH 4th, Cohen SP. Epidural injections for spinal pain: a systematic review and meta-analysis evaluating the "control" injections in randomized controlled trials. Anesthesiology. 2013 Oct;119(4):907-31. doi: 10.1097/ALN.0b013e31829c2ddd. PMID 24195874
- [Background] Blease C, Colloca L, Kaptchuk TJ. Are open-Label Placebos Ethical? Informed Consent and Ethical Equivocations. Bioethics. 2016 Jul;30(6):407-14. doi: 10.1111/bioe.12245. Epub 2016 Feb 3. PMID 26840547
- [Background] Bushnell MC, Ceko M, Low LA. Cognitive and emotional control of pain and its disruption in chronic pain. Nat Rev Neurosci. 2013 Jul;14(7):502-11. doi: 10.1038/nrn3516. Epub 2013 May 30. PMID 23719569
- [Background] Cherkin DC, Sherman KJ, Balderson BH, Cook AJ, Anderson ML, Hawkes RJ, Hansen KE, Turner JA. Effect of Mindfulness-Based Stress Reduction vs Cognitive Behavioral Therapy or Usual Care on Back Pain and Functional Limitations in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1240-9. doi: 10.1001/jama.2016.2323. PMID 27002445
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] Cohen SP, Argoff CE, Carragee EJ. Management of low back pain. BMJ. 2008 Dec 22;337:a2718. doi: 10.1136/bmj.a2718. No abstract available. PMID 19103627
- [Background] Colloca L, Petrovic P, Wager TD, Ingvar M, Benedetti F. How the number of learning trials affects placebo and nocebo responses. Pain. 2010 Nov;151(2):430-439. doi: 10.1016/j.pain.2010.08.007. PMID 20817355
- [Background] Delgado MR, Li J, Schiller D, Phelps EA. The role of the striatum in aversive learning and aversive prediction errors. Philos Trans R Soc Lond B Biol Sci. 2008 Dec 12;363(1511):3787-800. doi: 10.1098/rstb.2008.0161. PMID 18829426
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK; National Institutes of Health task force on research standards for chronic low back pain. Report of the National Institutes of Health task force on research standards for chronic low back pain. J Manipulative Physiol Ther. 2014 Sep;37(7):449-67. doi: 10.1016/j.jmpt.2014.07.006. Epub 2014 Aug 12. PMID 25127996
- [Background] Dimidjian S, Goodman SH, Felder JN, Gallop R, Brown AP, Beck A. Staying well during pregnancy and the postpartum: A pilot randomized trial of mindfulness-based cognitive therapy for the prevention of depressive relapse/recurrence. J Consult Clin Psychol. 2016 Feb;84(2):134-45. doi: 10.1037/ccp0000068. Epub 2015 Dec 14. PMID 26654212
- [Background] Dimidjian S, Hollon SD. How would we know if psychotherapy were harmful? Am Psychol. 2010 Jan;65(1):21-33. doi: 10.1037/a0017299. PMID 20063907
- [Background] Dimidjian S, Hollon SD, Dobson KS, Schmaling KB, Kohlenberg RJ, Addis ME, Gallop R, McGlinchey JB, Markley DK, Gollan JK, Atkins DC, Dunner DL, Jacobson NS. Randomized trial of behavioral activation, cognitive therapy, and antidepressant medication in the acute treatment of adults with major depression. J Consult Clin Psychol. 2006 Aug;74(4):658-70. doi: 10.1037/0022-006X.74.4.658. PMID 16881773
- [Background] Eldar E, Hauser TU, Dayan P, Dolan RJ. Striatal structure and function predict individual biases in learning to avoid pain. Proc Natl Acad Sci U S A. 2016 Apr 26;113(17):4812-7. doi: 10.1073/pnas.1519829113. Epub 2016 Apr 11. PMID 27071092
- [Background] Freburger JK, Holmes GM, Agans RP, Jackman AM, Darter JD, Wallace AS, Castel LD, Kalsbeek WD, Carey TS. The rising prevalence of chronic low back pain. Arch Intern Med. 2009 Feb 9;169(3):251-8. doi: 10.1001/archinternmed.2008.543. PMID 19204216
- [Background] Gatchel RJ, Peng YB, Peters ML, Fuchs PN, Turk DC. The biopsychosocial approach to chronic pain: scientific advances and future directions. Psychol Bull. 2007 Jul;133(4):581-624. doi: 10.1037/0033-2909.133.4.581. PMID 17592957
- [Background] Geuter S, Buchel C. Facilitation of pain in the human spinal cord by nocebo treatment. J Neurosci. 2013 Aug 21;33(34):13784-90. doi: 10.1523/JNEUROSCI.2191-13.2013. PMID 23966699
- [Background] Geuter S, Eippert F, Hindi Attar C, Buchel C. Cortical and subcortical responses to high and low effective placebo treatments. Neuroimage. 2013 Feb 15;67:227-36. doi: 10.1016/j.neuroimage.2012.11.029. Epub 2012 Nov 28. PMID 23201367
- [Background] Grace PM, Hutchinson MR, Maier SF, Watkins LR. Pathological pain and the neuroimmune interface. Nat Rev Immunol. 2014 Apr;14(4):217-31. doi: 10.1038/nri3621. Epub 2014 Feb 28. PMID 24577438
- [Background] Haake M, Muller HH, Schade-Brittinger C, Basler HD, Schafer H, Maier C, Endres HG, Trampisch HJ, Molsberger A. German Acupuncture Trials (GERAC) for chronic low back pain: randomized, multicenter, blinded, parallel-group trial with 3 groups. Arch Intern Med. 2007 Sep 24;167(17):1892-8. doi: 10.1001/archinte.167.17.1892. PMID 17893311
- [Background] Hashmi JA, Baliki MN, Huang L, Baria AT, Torbey S, Hermann KM, Schnitzer TJ, Apkarian AV. Shape shifting pain: chronification of back pain shifts brain representation from nociceptive to emotional circuits. Brain. 2013 Sep;136(Pt 9):2751-68. doi: 10.1093/brain/awt211. PMID 23983029
- [Background] Hashmi JA, Baria AT, Baliki MN, Huang L, Schnitzer TJ, Apkarian VA. Brain networks predicting placebo analgesia in a clinical trial for chronic back pain. Pain. 2012 Dec;153(12):2393-2402. doi: 10.1016/j.pain.2012.08.008. Epub 2012 Sep 15. PMID 22985900
- [Background] Hashmi JA, Baliki MN, Huang L, Parks EL, Chanda ML, Schnitzer T, Apkarian AV. Lidocaine patch (5%) is no more potent than placebo in treating chronic back pain when tested in a randomised double blind placebo controlled brain imaging study. Mol Pain. 2012 Apr 24;8:29. doi: 10.1186/1744-8069-8-29. PMID 22531485
- [Background] Hoffman BM, Papas RK, Chatkoff DK, Kerns RD. Meta-analysis of psychological interventions for chronic low back pain. Health Psychol. 2007 Jan;26(1):1-9. doi: 10.1037/0278-6133.26.1.1. PMID 17209691
- [Background] Hrobjartsson A, Gotzsche PC. Placebo interventions for all clinical conditions. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD003974. doi: 10.1002/14651858.CD003974.pub3. PMID 20091554
- [Background] Hsu MC, Schubiner H, Lumley MA, Stracks JS, Clauw DJ, Williams DA. Sustained pain reduction through affective self-awareness in fibromyalgia: a randomized controlled trial. J Gen Intern Med. 2010 Oct;25(10):1064-70. doi: 10.1007/s11606-010-1418-6. Epub 2010 Jun 8. PMID 20532650
- [Background] Hull SC, Colloca L, Avins A, Gordon NP, Somkin CP, Kaptchuk TJ, Miller FG. Patients' attitudes about the use of placebo treatments: telephone survey. BMJ. 2013 Jul 2;347:f3757. doi: 10.1136/bmj.f3757. PMID 23819963
- [Background] Irwin MR, Miller AH. Depressive disorders and immunity: 20 years of progress and discovery. Brain Behav Immun. 2007 May;21(4):374-83. doi: 10.1016/j.bbi.2007.01.010. Epub 2007 Mar 13. PMID 17360153
- [Background] Jensen MP, Ehde DM, Day MA. The Behavioral Activation and Inhibition Systems: Implications for Understanding and Treating Chronic Pain. J Pain. 2016 May;17(5):529.e1-529.e18. doi: 10.1016/j.jpain.2016.02.001. Epub 2016 Mar 24. PMID 27052644
- [Background] Kam-Hansen S, Jakubowski M, Kelley JM, Kirsch I, Hoaglin DC, Kaptchuk TJ, Burstein R. Altered placebo and drug labeling changes the outcome of episodic migraine attacks. Sci Transl Med. 2014 Jan 8;6(218):218ra5. doi: 10.1126/scitranslmed.3006175. PMID 24401940
- [Background] Kaptchuk TJ. The placebo effect in alternative medicine: can the performance of a healing ritual have clinical significance? Ann Intern Med. 2002 Jun 4;136(11):817-25. doi: 10.7326/0003-4819-136-11-200206040-00011. PMID 12044130
- [Background] Kaptchuk TJ, Friedlander E, Kelley JM, Sanchez MN, Kokkotou E, Singer JP, Kowalczykowski M, Miller FG, Kirsch I, Lembo AJ. Placebos without deception: a randomized controlled trial in irritable bowel syndrome. PLoS One. 2010 Dec 22;5(12):e15591. doi: 10.1371/journal.pone.0015591. PMID 21203519
- [Background] Kelley JM, Kaptchuk TJ, Cusin C, Lipkin S, Fava M. Open-label placebo for major depressive disorder: a pilot randomized controlled trial. Psychother Psychosom. 2012;81(5):312-4. doi: 10.1159/000337053. Epub 2012 Aug 1. No abstract available. PMID 22854752
- [Background] Koban L, Wager TD. Beyond conformity: Social influences on pain reports and physiology. Emotion. 2016 Feb;16(1):24-32. doi: 10.1037/emo0000087. Epub 2015 Aug 31. PMID 26322566
- [Background] Kregel J, Meeus M, Malfliet A, Dolphens M, Danneels L, Nijs J, Cagnie B. Structural and functional brain abnormalities in chronic low back pain: A systematic review. Semin Arthritis Rheum. 2015 Oct;45(2):229-37. doi: 10.1016/j.semarthrit.2015.05.002. Epub 2015 May 16. PMID 26092329
- [Background] Lee M, Manders TR, Eberle SE, Su C, D'amour J, Yang R, Lin HY, Deisseroth K, Froemke RC, Wang J. Activation of corticostriatal circuitry relieves chronic neuropathic pain. J Neurosci. 2015 Apr 1;35(13):5247-59. doi: 10.1523/JNEUROSCI.3494-14.2015. PMID 25834050
- [Background] Manchikanti L, Pampati V, Falco FJ, Hirsch JA. Growth of spinal interventional pain management techniques: analysis of utilization trends and Medicare expenditures 2000 to 2008. Spine (Phila Pa 1976). 2013 Jan 15;38(2):157-68. doi: 10.1097/BRS.0b013e318267f463. PMID 22781007
- [Background] Miller FG, Kaptchuk TJ. The power of context: reconceptualizing the placebo effect. J R Soc Med. 2008 May;101(5):222-5. doi: 10.1258/jrsm.2008.070466. No abstract available. PMID 18463276
- [Background] Moore RC, Depp CA, Wetherell JL, Lenze EJ. Ecological momentary assessment versus standard assessment instruments for measuring mindfulness, depressed mood, and anxiety among older adults. J Psychiatr Res. 2016 Apr;75:116-23. doi: 10.1016/j.jpsychires.2016.01.011. Epub 2016 Jan 22. PMID 26851494
- [Background] Muller M, Kamping S, Benrath J, Skowronek H, Schmitz J, Klinger R, Flor H. Treatment history and placebo responses to experimental and clinical pain in chronic pain patients. Eur J Pain. 2016 Oct;20(9):1530-41. doi: 10.1002/ejp.877. Epub 2016 Apr 7. PMID 27062187
- [Background] Ortiz R, Chandros Hull S, Colloca L. Patient attitudes about the clinical use of placebo: qualitative perspectives from a telephone survey. BMJ Open. 2016 Apr 4;6(4):e011012. doi: 10.1136/bmjopen-2015-011012. PMID 27044586
- [Background] Pedersen LM, Schistad E, Jacobsen LM, Roe C, Gjerstad J. Serum levels of the pro-inflammatory interleukins 6 (IL-6) and -8 (IL-8) in patients with lumbar radicular pain due to disc herniation: A 12-month prospective study. Brain Behav Immun. 2015 May;46:132-6. doi: 10.1016/j.bbi.2015.01.008. Epub 2015 Jan 31. PMID 25653193
- [Background] Roy M, Shohamy D, Daw N, Jepma M, Wimmer GE, Wager TD. Representation of aversive prediction errors in the human periaqueductal gray. Nat Neurosci. 2014 Nov;17(11):1607-12. doi: 10.1038/nn.3832. Epub 2014 Oct 5. PMID 25282614
- [Background] Schafer SM, Colloca L, Wager TD. Conditioned placebo analgesia persists when subjects know they are receiving a placebo. J Pain. 2015 May;16(5):412-20. doi: 10.1016/j.jpain.2014.12.008. Epub 2015 Jan 22. PMID 25617812
- [Background] Schistad EI, Espeland A, Pedersen LM, Sandvik L, Gjerstad J, Roe C. Association between baseline IL-6 and 1-year recovery in lumbar radicular pain. Eur J Pain. 2014 Nov;18(10):1394-401. doi: 10.1002/j.1532-2149.2014.502.x. Epub 2014 Apr 2. PMID 24692238
- [Background] Schwartz N, Temkin P, Jurado S, Lim BK, Heifets BD, Polepalli JS, Malenka RC. Chronic pain. Decreased motivation during chronic pain requires long-term depression in the nucleus accumbens. Science. 2014 Aug 1;345(6196):535-42. doi: 10.1126/science.1253994. PMID 25082697
- [Background] Seminowicz DA, Wideman TH, Naso L, Hatami-Khoroushahi Z, Fallatah S, Ware MA, Jarzem P, Bushnell MC, Shir Y, Ouellet JA, Stone LS. Effective treatment of chronic low back pain in humans reverses abnormal brain anatomy and function. J Neurosci. 2011 May 18;31(20):7540-50. doi: 10.1523/JNEUROSCI.5280-10.2011. PMID 21593339
- [Background] Seymour B, O'Doherty JP, Koltzenburg M, Wiech K, Frackowiak R, Friston K, Dolan R. Opponent appetitive-aversive neural processes underlie predictive learning of pain relief. Nat Neurosci. 2005 Sep;8(9):1234-40. doi: 10.1038/nn1527. Epub 2005 Aug 21. PMID 16116445
- [Background] Shallcross AJ, Gross JJ, Visvanathan PD, Kumar N, Palfrey A, Ford BQ, Dimidjian S, Shirk S, Holm-Denoma J, Goode KM, Cox E, Chaplin W, Mauss IB. Relapse prevention in major depressive disorder: Mindfulness-based cognitive therapy versus an active control condition. J Consult Clin Psychol. 2015 Oct;83(5):964-75. doi: 10.1037/ccp0000050. Epub 2015 Aug 10. PMID 26371618
- [Background] Shpaner M, Kelly C, Lieberman G, Perelman H, Davis M, Keefe FJ, Naylor MR. Unlearning chronic pain: A randomized controlled trial to investigate changes in intrinsic brain connectivity following Cognitive Behavioral Therapy. Neuroimage Clin. 2014 Jul 23;5:365-76. doi: 10.1016/j.nicl.2014.07.008. eCollection 2014. PMID 26958466
- [Background] Tilburt JC, Emanuel EJ, Kaptchuk TJ, Curlin FA, Miller FG. Prescribing "placebo treatments": results of national survey of US internists and rheumatologists. BMJ. 2008 Oct 23;337:a1938. doi: 10.1136/bmj.a1938. PMID 18948346
- [Background] Tuttle AH, Tohyama S, Ramsay T, Kimmelman J, Schweinhardt P, Bennett GJ, Mogil JS. Increasing placebo responses over time in U.S. clinical trials of neuropathic pain. Pain. 2015 Dec;156(12):2616-2626. doi: 10.1097/j.pain.0000000000000333. PMID 26307858
- [Background] Vachon-Presseau E, Tetreault P, Petre B, Huang L, Berger SE, Torbey S, Baria AT, Mansour AR, Hashmi JA, Griffith JW, Comasco E, Schnitzer TJ, Baliki MN, Apkarian AV. Corticolimbic anatomical characteristics predetermine risk for chronic pain. Brain. 2016 Jul;139(Pt 7):1958-70. doi: 10.1093/brain/aww100. Epub 2016 May 5. PMID 27190016
- [Background] Vlaev I, Seymour B, Chater N, Winston JS, Yoshida W, Wright N, Symmonds M, Dolan R. Prices need no preferences: social trends determine decisions in experimental markets for pain relief. Health Psychol. 2014 Jan;33(1):66-76. doi: 10.1037/a0030372. Epub 2012 Nov 12. PMID 23148449
- [Background] Vlaev I, Seymour B, Dolan RJ, Chater N. The price of pain and the value of suffering. Psychol Sci. 2009 Mar;20(3):309-17. doi: 10.1111/j.1467-9280.2009.02304.x. Epub 2009 Feb 23. PMID 19254237
- [Background] Wager TD, Atlas LY. The neuroscience of placebo effects: connecting context, learning and health. Nat Rev Neurosci. 2015 Jul;16(7):403-18. doi: 10.1038/nrn3976. PMID 26087681
- [Background] Wager TD, Atlas LY, Leotti LA, Rilling JK. Predicting individual differences in placebo analgesia: contributions of brain activity during anticipation and pain experience. J Neurosci. 2011 Jan 12;31(2):439-52. doi: 10.1523/JNEUROSCI.3420-10.2011. PMID 21228154
- [Background] Wager TD, Atlas LY, Lindquist MA, Roy M, Woo CW, Kross E. An fMRI-based neurologic signature of physical pain. N Engl J Med. 2013 Apr 11;368(15):1388-97. doi: 10.1056/NEJMoa1204471. PMID 23574118
- [Background] Wager TD, Rilling JK, Smith EE, Sokolik A, Casey KL, Davidson RJ, Kosslyn SM, Rose RM, Cohen JD. Placebo-induced changes in FMRI in the anticipation and experience of pain. Science. 2004 Feb 20;303(5661):1162-7. doi: 10.1126/science.1093065. PMID 14976306
- [Background] Winston JS, Vlaev I, Seymour B, Chater N, Dolan RJ. Relative valuation of pain in human orbitofrontal cortex. J Neurosci. 2014 Oct 29;34(44):14526-35. doi: 10.1523/JNEUROSCI.1706-14.2014. PMID 25355207
- [Derived] Ashar YK, Sun M, Knight K, Flood TF, Anderson Z, Kaptchuk TJ, Wager TD. Open-Label Placebo Injection for Chronic Back Pain With Functional Neuroimaging: A Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2432427. doi: 10.1001/jamanetworkopen.2024.32427. PMID 39259542
- [Derived] Ashar YK, Gordon A, Schubiner H, Uipi C, Knight K, Anderson Z, Carlisle J, Polisky L, Geuter S, Flood TF, Kragel PA, Dimidjian S, Lumley MA, Wager TD. Effect of Pain Reprocessing Therapy vs Placebo and Usual Care for Patients With Chronic Back Pain: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Jan 1;79(1):13-23. doi: 10.1001/jamapsychiatry.2021.2669. PMID 34586357

RESULTS

PARTICIPANT FLOW:
Groups:
- Pain Reprocessing Therapy (PRT): Received psychological treatment
- Placebo: Open-label placebo
- Usual Care: Continue usual care
Period: Overall Study
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Started | 50 | 51 | 50
Completed | 44 | 44 | 47
Not Completed | 6 | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care | Total
Number analyzed (Participants) | 50 | 51 | 50 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (16.2) | 39.4 (14.9) | 41.3 (15.9) | 41.1 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 27 | 81
  Male | 21 | 26 | 23 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 50 | 49 | 48 | 147
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 46 | 45 | 43 | 134
  More than one race | 1 | 2 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory-Short Form (BPI-SF)
Description: 1-week average pain intensity, 0 - 10 numerical rating scale, where a higher score indicates more pain.
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pain Reprocessing Therapy (PRT): Psychological treatment
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
units on a scale | 1.18 (1.24) | 2.84 (1.64) | 3.13 (1.45)

2. Secondary Outcome: Positive Affect Scale Short Form (PANAS-SF)
Description: Questionnaire to rate positive affect, scores range from 5 - 25, a higher score means stronger affect
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
score on a scale | 17.89 (3.38) | 15.20 (5.60) | 14.98 (3.50)

3. Secondary Outcome: PROMIS- Depression
Description: Questionnaire measuring depression (8 items). Scores range from 8-32. A higher score indicates higher levels of depressive symptoms
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
score on a scale | 12.23 (4.94) | 11.75 (4.05) | 11.81 (4.45)

4. Secondary Outcome: Tampa Scale of Kinesiophobia (TSK)
Description: Questionnaire used to assess the subjective rating of kinesiophobia or fear of movement. Scores range from 11-44 with higher scores indicating greater fear of pain, movement, and injury.
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
score on a scale | 16.41 (5.37) | 22.16 (4.94) | 22.51 (6.30)

5. Secondary Outcome: Pain Catastrophizing Questionnaire (PCS)
Description: Questionnaire used to help quantify an individual's pain experience. Measured 0-52. A higher score means a higher level of catastrophizing.
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
score on a scale | 8.30 (3.04) | 7.70 (2.44) | 8.19 (2.75)

6. Secondary Outcome: Timeline Follow-Back Measure for Alcohol (TLFB)
Description: Questionnaire used to assess daily drinking (number of drinks consumed over past two weeks)
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: Drinks
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
Drinks | 11.63 (10.83) | 12.88 (14.30) | 8.02 (10.63)

7. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Post-treatment-only outcome measure depicting a patient's subjective rating of overall improvement. Score ranges from 1-7 with a higher score indicating a higher level of change and improvement
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
score on a scale | 6.14 (0.88) | 3.61 (1.62) | 2.06 (1.45)

8. Secondary Outcome: Treatment Satisfaction Questionnaire
Description: Post-treatment-only outcome measure depicting the patient's satisfaction with the treatment. Measured 0 - 100. A higher score means higher satisfaction with treatment/
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
score on a scale | 92.40 (8.01) | 57.61 (23.05) | 36.86 (23.01)

9. Secondary Outcome: Oswestry Disability Index
Description: Back pain disability questionnaire measured on a scale of 0-100. A higher score indicates a higher severity of disability.
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
score on a scale | 10.14 (10.63) | 19.00 (11.07) | 20.68 (10.68)

10. Secondary Outcome: Negative Affect Scale Short Form (PANAS-SF)
Description: Questionnaire to rate negative affect, scores range from 5 - 25, with a higher score meaning a stronger negative affect
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
score on a scale | 8.30 (3.04) | 7.70 (2.44) | 8.19 (2.75)

11. Secondary Outcome: PROMIS Anger
Description: Questionnaire measuring anger (5 items) with a score range of 5-25. Higher scores indicate a higher severity of anger.
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
score on a scale | 9.52 (3.91) | 9.89 (3.81) | 10.45 (3.86)

12. Secondary Outcome: PROMIS Sleep
Description: Questionnaire measuring sleep disturbance (8 items). Scores range from 8-40. Higher scores indicate higher levels of sleep disturbance
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
score on a scale | 17.73 (6.75) | 20.50 (6.17) | 20.89 (6.02)

13. Secondary Outcome: PROMIS Anxiety
Description: Questionnaire measuring anxiety (8 items). Scores range from 8-40 with a higher score meaning more severe levels of fear, anxious misery, hyperarousal, and somatic symptoms related to arousal.
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
score on a scale | 15.02 (6.16) | 13.89 (5.78) | 14.11 (6.99)

14. Secondary Outcome: Timeline Follow-Back Measure for Opioid Use (TLFB)
Description: Questionnaire used to assess daily opioid use (number of pills consumed over past two weeks)
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: Opioid pills
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
Opioid pills | 1.29 (4.50) | 0.36 (2.11) | 1.77 (8.99)

15. Secondary Outcome: Timeline Follow-Back Measure for Cannabis (TLFB)
Description: Questionnaire used to assess daily cannabis use (number of grams consumed over past two weeks)
Time Frame: At post-treatment fMRI session, approximately 1 month after randomization
Population: all available participants analyzed
Measure: Mean (Standard Deviation); unit: Grams of cannabis
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
Number analyzed (Participants) | 44 | 44 | 47
Grams of cannabis | 6.76 (25.32) | 3.31 (6.72) | 1.49 (3.20)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through completion of the post-treatment fMRI session, an average of 1.5 months after enrollment.
Description: Adverse events were recorded when participants spontaneously reported them to study personnel.
Arm/Group | Pain Reprocessing Therapy (PRT) | Placebo | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/51 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT03294148/Prot_SAP_004.pdf
  • Informed Consent Form: Placebo (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT03294148/ICF_005.pdf
  • Informed Consent Form: Control (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT03294148/ICF_006.pdf
  • Informed Consent Form: Psychotherapy (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT03294148/ICF_007.pdf